CLINICAL TRIAL: NCT03770845
Title: Nutritional Assessment in Idiopathic Pulmonary Fibrosis: a Pilot Study
Brief Title: Nutritional Assessment in Idiopathic Pulmonary Fibrosis
Acronym: NUTRIPF
Status: Completed | Type: Observational
Sponsor: San Gerardo Hospital (Other)
Responsible Party: Principal Investigator, Paola Faverio, Principal Investigator, San Gerardo Hospital
Other Study IDs: NUTRIPF
Record Dates: First submitted 2018-12-06; First posted 2018-12-10 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: nutritional status; vitamin D
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In recent years nutritional status assumed increasing importance in the evaluation of chronic respiratory diseases, considering that their clinical course is often characterized by a progressive loss of weight and reduction of muscle mass.In regards to Idiopathic Pulmonary Fibrosis (IPF), to date there are no studies that fully assessed the nutritional status of patients, nor the impact of the introduction of specific anti-fibrotic agents on the nutritional status of these patients.

Aim of this study is to assess the nutritional status of patients with IPF at the time of diagnosis and the impact of the introduction of specific anti-fibrotic agents, pirfenidone or nintedanib, on the nutritional status itself.

DETAILED DESCRIPTION:
Preliminary studies on Idiopathic Pulmonary Fibrosis (IPF) seem to suggest that nutritional status has an impact on clinical outcomes, as already demonstrated in COPD. However, few data regarding this subject are available for patients with IPF.

Primary aim of this study is to assess the nutritional status of patients diagnosed with mild to moderate IPF at the time of disease diagnosis. To do so, the investigators assess the prevalence of nutritional disorders at baseline through nutritional scores evaluated with specific questionnaires and through the identification of the following metabolic phenotypes (based on those previously applied in COPD): cachexia, sarcopenia, normal nutritional status, obesity, sarcopenic obesity.

Secondary aims of this study are:

* the evaluation of the impact of the introduction of an anti-fibrotic pharmacological agent (pirfenidone or nintedanib) on the nutritional status of patients (modification of metabolic phenotypes and nutritional scores) evaluated at 6 months from the initiation of antifibrotic therapy.
* the assessment of calcium and vitamin D metabolism, by blood sampling, in patients diagnosed with mild to moderate IPF at the time of disease diagnosis and at 6 months from the initiation of antifibrotic therapy.

ELIGIBILITY:
Inclusion Criteria:

* age greater than or equal to 18 years;
* diagnosis of IPF according to the ATS / ERS 2011 guidelines with multidisciplinary discussion

Exclusion Criteria:

* severe renal failure, defined as a GFR (glomerular filtration rate) lower than 30ml / min;
* NYHA class IV;
* severe liver failure, defined as Child-Pugh score class C;
* active solid or haematological neoplasms;
* having already received (currently or in the past) therapy with pirfenidone or nintedanib;
* inability to walk without help;
* need for oxygen therapy at rest;
* participation in other interventional experimental protocols with use of a medicinal product.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a diagnosis of mild to moderate Idiopathic Pulmonary Fibrosis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
BMI (body mass index) | baseline (IPF diagnosis)
  kg/m2
FFMI (fat free mass index) | baseline (IPF diagnosis)
  kg/m2
SMI (skeletal muscle mass index) | baseline (IPF diagnosis)
  kg/m2
BFMI (body fat mass index) | baseline (IPF diagnosis)
  kg/m2
Hand Grip | baseline (IPF diagnosis)
  kg
Abdominal circumference | baseline (IPF diagnosis)
  cm
Malnutrition Universal Screening Tool (MUST) Screening Tool (MUST) | baseline (IPF diagnosis)
  questionnaire score: score 0 = low risk of malnutrition; score 1 = medium risk of malnutrition; score equal or higher than 2 = high risk of malnutrition
Mini Nutritional Assessment (MNA) | baseline (IPF diagnosis)
  questionnaire score (maximum score 30): total score > 23.5 = normal nutritional status; total score < 23.5 = inadequate nutritional status

SECONDARY OUTCOMES:
BMI (body mass index) | 6 months after baseline
  kg/m2
FFMI (fat free mass index) | 6 months after baseline
  kg/m2
SMI (skeletal muscle mass index) | 6 months after baseline
  kg/m2
BFMI (body fat mass index) | 6 months after baseline
  kg/m2
Hand Grip | 6 months after baseline
  kg
Abdominal circumference | 6 months after baseline
  cm
Malnutrition Universal Screening Tool (MUST) | 6 months after baseline
  questionnaire score: score 0 = low risk of malnutrition; score 1 = medium risk of malnutrition; score equal or higher than 2 = high risk of malnutrition
Mini Nutritional Assessment (MNA) | 6 months after baseline
  questionnaire score (maximum score 30): total score > 23.5 = normal nutritional status; total score < 23.5 = inadequate nutritional status
plasma calcium | baseline (IPF diagnosis) and 6 months after baseline
  calcium level in plasma
plasma vitamin D | baseline (IPF diagnosis) and 6 months after baseline
  vitamin D level in plasma

CONTACTS AND LOCATIONS:
Locations (9):
- Italy (9):
  - INRCA Casatenovo, Casatenovo, Lecco
  - San Gerardo Hospital, Monza, MB
  - G. Salvini Hospital, Garbagnate Milanese, Milano
  - Ospedale di Circolo, Busto Arsizio, Varese
  - Ospedale SS. Annunziata, Chieti
  - San Martino Hospital, Genova
  - San Giuseppe Hospital, Milan
  - San Paolo and San Carlo Hospital, Milan
  - Ospedale Maggiore Novara, Novara

IPD SHARING:
Plan to Share IPD: No